CLINICAL TRIAL: NCT03605498
Title: An Investigation of Novel Technology to Bring Genomic Analysis to the Patient Bedside to Systematically Track and Report on ESKAPE Bacterial Transmission in Today's Operating Room Environments
Brief Title: OR PathTrac (Tracking Intra-operative Bacterial Transmission)
Status: Completed | Type: Observational
Sponsor: Sundara Reddy (Other)
Collaborators: B. Braun Medical Inc. (Industry); RDB Bioinformatics (Industry)
Responsible Party: Sponsor-Investigator, Sundara Reddy, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201705826
Record Dates: First submitted 2018-06-08; First posted 2018-07-30 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The bacterial cultures can be kept and analyzed at a later date to determine how they have transformed into antibiotic resistant organisms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthcare-associated infections occur frequently and are associated with patient harm. These infections are becoming more difficult to treat due to antibiotic resistance. It is important that healthcare facilities take the steps necessary to prevent the spread of resistant bacteria between patients.

DETAILED DESCRIPTION:
Two patients undergoing sedation in a randomly selected operating room will be evaluated in a serial manner in order to detect transmission of pathogenic bacteria. Patient care will not change due to their participation in this study; the patients will undergo sedation and surgery according to usual practice. This study involves taking microbiology cultures from various places in the operating room before and after each procedure. Cultures will also be taken from the two patients after they are asleep and from their intravenous tubing. From both patients anesthesiologist, surgeon and their surgical team, cRNA, and nursing staff will also have cultures obtained. Each cultures will be de-identified and given a study ID number before transport to the research laboratory for microbiological assay. The patient's medical record will be reviewed for 30 days after surgery to surveil for documentation of a potential hospital acquired infection.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Require peripheral intravenous and/or central venous catheter placement
* Undergoing gynecology/oncology, colorectal, open vascular, total joint or cardiovascular procedures.

Exclusion Criteria:

* Less than 18 years of age
* Does not require peripheral intravenous and/or central venous catheter placement
* Patient refusal to participate
* Incarceration

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be surgical patients requiring peripheral intravenous and/or central venous catheter access and undergoing gynecology/oncology, colorectal, open vascular, total joint or cardiovascular procedures.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Identify transmission dynamics of pathogenic bacteria (i.e. Staph aureus). | Intraoperative period
  Focus on how Staph aureus is transmitted in the operating room by identifying key areas of origin.
Intraoperative clonal transmission of Staph aureus. | Intraoperative period
  Monitor locations throughout the operating room to document clonal transmission from the area of origin.
Identify the modes of transmission of pathogenic bacteria ((i.e. Staph aureus). | Intraoperative period
  If transmission of Staph aureus from the site of origin to another site in the operating room arena is documented, identify the modes of transmission.

SECONDARY OUTCOMES:
Monitor for post operative healthcare associated infections. | Up to 30 days following surgery
  Monitor for the presence or absence of healthcare associated infection after undergoing an operative procedure.
Surveil for molecular links between pathogenic organisms. | Up to 30 days following surgery
  Seek to identify molecular links between causative organisms of infection and bacteria found in the operating room at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sundara Reddy, MBBS, FRCA, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal

REFERENCES:
- [Background] Vogel TR, Dombrovskiy VY, Lowry SF. Impact of infectious complications after elective surgery on hospital readmission and late deaths in the U.S. Medicare population. Surg Infect (Larchmt). 2012 Oct;13(5):307-11. doi: 10.1089/sur.2012.116. Epub 2012 Oct 19. PMID 23082877
- [Background] Koff MD, Brown JR, Marshall EJ, O'Malley AJ, Jensen JT, Heard SO, Longtine K, O'Neill M, Longtine J, Houston D, Robison C, Moulton E, Patel HM, Loftus RW. Frequency of Hand Decontamination of Intraoperative Providers and Reduction of Postoperative Healthcare-Associated Infections: A Randomized Clinical Trial of a Novel Hand Hygiene System. Infect Control Hosp Epidemiol. 2016 Aug;37(8):888-895. doi: 10.1017/ice.2016.106. Epub 2016 Jun 7. PMID 27267310
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] World Health Organization. Antimicrobial Resistance. Global Report on Surveillance, WHO. 2014
- [Background] German RR, Lee LM, Horan JM, Milstein RL, Pertowski CA, Waller MN; Guidelines Working Group Centers for Disease Control and Prevention (CDC). Updated guidelines for evaluating public health surveillance systems: recommendations from the Guidelines Working Group. MMWR Recomm Rep. 2001 Jul 27;50(RR-13):1-35; quiz CE1-7. PMID 18634202
- [Background] Boucher HW, Talbot GH, Bradley JS, Edwards JE, Gilbert D, Rice LB, Scheld M, Spellberg B, Bartlett J. Bad bugs, no drugs: no ESKAPE! An update from the Infectious Diseases Society of America. Clin Infect Dis. 2009 Jan 1;48(1):1-12. doi: 10.1086/595011. PMID 19035777
- [Background] Loftus RW, Koff MD, Burchman CC, Schwartzman JD, Thorum V, Read ME, Wood TA, Beach ML. Transmission of pathogenic bacterial organisms in the anesthesia work area. Anesthesiology. 2008 Sep;109(3):399-407. doi: 10.1097/ALN.0b013e318182c855. PMID 18719437
- [Background] Loftus RW, Brown JR, Koff MD, Reddy S, Heard SO, Patel HM, Fernandez PG, Beach ML, Corwin HL, Jensen JT, Kispert D, Huysman B, Dodds TM, Ruoff KL, Yeager MP. Multiple reservoirs contribute to intraoperative bacterial transmission. Anesth Analg. 2012 Jun;114(6):1236-48. doi: 10.1213/ANE.0b013e31824970a2. Epub 2012 Mar 30. PMID 22467892
- [Background] Loftus RW, Koff MD, Brown JR, Patel HM, Jensen JT, Reddy S, Ruoff KL, Heard SO, Yeager MP, Dodds TM. The epidemiology of Staphylococcus aureus transmission in the anesthesia work area. Anesth Analg. 2015 Apr;120(4):807-18. doi: 10.1213/ANE.0b013e3182a8c16a. PMID 24937345
- [Background] Loftus RW, Koff MD, Brown JR, Patel HM, Jensen JT, Reddy S, Ruoff KL, Heard SO, Yeager MP, Dodds TM. The dynamics of Enterococcus transmission from bacterial reservoirs commonly encountered by anesthesia providers. Anesth Analg. 2015 Apr;120(4):827-36. doi: 10.1213/ANE.0000000000000123. PMID 24937346
- [Background] Loftus RW, Brown JR, Patel HM, Koff MD, Jensen JT, Reddy S, Ruoff KL, Heard SO, Dodds TM, Beach ML, Yeager MP. Transmission dynamics of gram-negative bacterial pathogens in the anesthesia work area. Anesth Analg. 2015 Apr;120(4):819-26. doi: 10.1213/ANE.0000000000000626. PMID 25790209
- [Background] Mabit C, Marcheix PS, Mounier M, Dijoux P, Pestourie N, Bonnevialle P, Bonnomet F; French Society of Orthopaedic Surgery, Traumatology (SOFCOT). Impact of a surgical site infection (SSI) surveillance program in orthopedics and traumatology. Orthop Traumatol Surg Res. 2012 Oct;98(6):690-5. doi: 10.1016/j.otsr.2012.08.001. Epub 2012 Sep 15. PMID 22986014
- [Background] Loftus RW, Muffly MK, Brown JR, Beach ML, Koff MD, Corwin HL, Surgenor SD, Kirkland KB, Yeager MP. Hand contamination of anesthesia providers is an important risk factor for intraoperative bacterial transmission. Anesth Analg. 2011 Jan;112(1):98-105. doi: 10.1213/ANE.0b013e3181e7ce18. Epub 2010 Aug 4. PMID 20686007
- [Background] Loftus RW, Patel HM, Huysman BC, Kispert DP, Koff MD, Gallagher JD, Jensen JT, Rowlands J, Reddy S, Dodds TM, Yeager MP, Ruoff KL, Surgenor SD, Brown JR. Prevention of intravenous bacterial injection from health care provider hands: the importance of catheter design and handling. Anesth Analg. 2012 Nov;115(5):1109-19. doi: 10.1213/ANE.0b013e31826a1016. Epub 2012 Oct 9. PMID 23051883
- [Background] Loftus RW, Brindeiro BS, Kispert DP, Patel HM, Koff MD, Jensen JT, Dodds TM, Yeager MP, Ruoff KL, Gallagher JD, Beach ML, Brown JR. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a passive catheter care system. Anesth Analg. 2012 Dec;115(6):1315-23. doi: 10.1213/ANE.0b013e31826d2aa4. Epub 2012 Nov 9. PMID 23144441
- [Background] Rowlands J, Yeager MP, Beach M, Patel HM, Huysman BC, Loftus RW. Video observation to map hand contact and bacterial transmission in operating rooms. Am J Infect Control. 2014 Jul;42(7):698-701. doi: 10.1016/j.ajic.2014.02.021. PMID 24969122
- [Background] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154
- [Background] Koff MD, Corwin HL, Beach ML, Surgenor SD, Loftus RW. Reduction in ventilator associated pneumonia in a mixed intensive care unit after initiation of a novel hand hygiene program. J Crit Care. 2011 Oct;26(5):489-495. doi: 10.1016/j.jcrc.2010.12.013. Epub 2011 Mar 24. PMID 21439767
- [Background] Edwards JR, Peterson KD, Mu Y, Banerjee S, Allen-Bridson K, Morrell G, Dudeck MA, Pollock DA, Horan TC. National Healthcare Safety Network (NHSN) report: data summary for 2006 through 2008, issued December 2009. Am J Infect Control. 2009 Dec;37(10):783-805. doi: 10.1016/j.ajic.2009.10.001. No abstract available. PMID 20004811
- [Background] Zerbino DR, Birney E. Velvet: algorithms for de novo short read assembly using de Bruijn graphs. Genome Res. 2008 May;18(5):821-9. doi: 10.1101/gr.074492.107. Epub 2008 Mar 18. PMID 18349386
- [Background] Perdiz LB, Yokoe DS, Furtado GH, Medeiros EAS. Impact of an Automated Surveillance to Detect Surgical-Site Infections in Patients Undergoing Total Hip and Knee Arthroplasty in Brazil. Infect Control Hosp Epidemiol. 2016 Aug;37(8):991-993. doi: 10.1017/ice.2016.86. Epub 2016 Apr 13. PMID 27072598
- [Background] Cheadle WG. Risk factors for surgical site infection. Surg Infect (Larchmt). 2006;7 Suppl 1:S7-11. doi: 10.1089/sur.2006.7.s1-7. PMID 16834549
- [Background] Owens CD, Stoessel K. Surgical site infections: epidemiology, microbiology and prevention. J Hosp Infect. 2008 Nov;70 Suppl 2:3-10. doi: 10.1016/S0195-6701(08)60017-1. PMID 19022115
- [Background] Qureshi ZA, Paterson DL, Pakstis DL, Adams-Haduch JM, Sandkovsky G, Sordillo E, Polsky B, Peleg AY, Bhussar MK, Doi Y. Risk factors and outcome of extended-spectrum beta-lactamase-producing Enterobacter cloacae bloodstream infections. Int J Antimicrob Agents. 2011 Jan;37(1):26-32. doi: 10.1016/j.ijantimicag.2010.09.009. Epub 2010 Nov 13. PMID 21075605
- [Background] Paryavi E, Stall A, Gupta R, Scharfstein DO, Castillo RC, Zadnik M, Hui E, O'Toole RV. Predictive model for surgical site infection risk after surgery for high-energy lower-extremity fractures: development of the risk of infection in orthopedic trauma surgery score. J Trauma Acute Care Surg. 2013 Jun;74(6):1521-7. doi: 10.1097/TA.0b013e318292158d. PMID 23694882
- [Background] Arnold C. Outbreak Breakthrough: Using Whole-Genome Sequencing to Control Hospital Infection. Environ Health Perspect. 2015 Nov;123(11):A281-6. doi: 10.1289/ehp.123-A281. No abstract available. PMID 26523889
- [Background] Rupp ME, Fitzgerald T, Puumala S, Anderson JR, Craig R, Iwen PC, Jourdan D, Keuchel J, Marion N, Peterson D, Sholtz L, Smith V. Prospective, controlled, cross-over trial of alcohol-based hand gel in critical care units. Infect Control Hosp Epidemiol. 2008 Jan;29(1):8-15. doi: 10.1086/524333. PMID 18171181
- [Background] Moureau NL, Flynn J. Disinfection of Needleless Connector Hubs: Clinical Evidence Systematic Review. Nurs Res Pract. 2015;2015:796762. doi: 10.1155/2015/796762. Epub 2015 May 14. PMID 26075093
- [Background] Schweizer ML, Chiang HY, Septimus E, Moody J, Braun B, Hafner J, Ward MA, Hickok J, Perencevich EN, Diekema DJ, Richards CL, Cavanaugh JE, Perlin JB, Herwaldt LA. Association of a bundled intervention with surgical site infections among patients undergoing cardiac, hip, or knee surgery. JAMA. 2015 Jun 2;313(21):2162-71. doi: 10.1001/jama.2015.5387. PMID 26034956
- [Background] Phillips M, Rosenberg A, Shopsin B, Cuff G, Skeete F, Foti A, Kraemer K, Inglima K, Press R, Bosco J. Preventing surgical site infections: a randomized, open-label trial of nasal mupirocin ointment and nasal povidone-iodine solution. Infect Control Hosp Epidemiol. 2014 Jul;35(7):826-32. doi: 10.1086/676872. Epub 2014 May 21. PMID 24915210
- [Background] Bode LG, Kluytmans JA, Wertheim HF, Bogaers D, Vandenbroucke-Grauls CM, Roosendaal R, Troelstra A, Box AT, Voss A, van der Tweel I, van Belkum A, Verbrugh HA, Vos MC. Preventing surgical-site infections in nasal carriers of Staphylococcus aureus. N Engl J Med. 2010 Jan 7;362(1):9-17. doi: 10.1056/NEJMoa0808939. PMID 20054045
- [Background] Konvalinka A, Errett L, Fong IW. Impact of treating Staphylococcus aureus nasal carriers on wound infections in cardiac surgery. J Hosp Infect. 2006 Oct;64(2):162-8. doi: 10.1016/j.jhin.2006.06.010. Epub 2006 Aug 23. PMID 16930768
- [Background] Chen YQ, Hu C, Wang Y. Attributable risk function in the proportional hazards model for censored time-to-event. Biostatistics. 2006 Oct;7(4):515-29. doi: 10.1093/biostatistics/kxj023. Epub 2006 Feb 14. PMID 16478758
- [Background] Mehrotra DV, Li X, Liu J, Lu K. Analysis of longitudinal clinical trials with missing data using multiple imputation in conjunction with robust regression. Biometrics. 2012 Dec;68(4):1250-9. doi: 10.1111/j.1541-0420.2012.01780.x. Epub 2012 Sep 20. PMID 22994905
- [Background] Carpenter J, Pocock S, Lamm CJ. Coping with missing data in clinical trials: a model-based approach applied to asthma trials. Stat Med. 2002 Apr 30;21(8):1043-66. doi: 10.1002/sim.1065. PMID 11933033
- [Background] Raudenbush SW. Hierarchical Linear Models: Applications and Data Analysis Methods. Newbury Park, CA: Sage; 2002.
- [Background] Wikler M, Cockerill F, Craig W, Dudley M, Eliopoulos G, Hecht P, Hindler J, Low D, Sheehan D, Tenover F, Turnidge J, Weinstein M, Zimmer B. Clinical and Laboratory Standards Institute: Performance Standards for Antimicrobial Disk Susceptibility Tests; Approved Standard-9th 10th edition. 2009, Wayne, PA, Clinical and Laboratory Standards Institute, 2006, pp M2 M02-A9A10